CLINICAL TRIAL: NCT02791477
Title: Functional Results With Attune Fixed Bearing Posterior Stabilized Knee Arthroplasty
Brief Title: Functional Results With Attune Fixed Bearing Posterior Stabilized Knee Arthroplasty (A-16)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Attune 2016
Record Dates: First submitted 2016-05-11; First posted 2016-06-06 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Knee Arthroplasty
Keywords: Attune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Attune FB PS (Other): Attune FB PS knee arthroplasty
  Interventions: Device: Attune FB PS knee arthroplasty

INTERVENTIONS:
Device: Attune FB PS knee arthroplasty

SUMMARY:
Functional results with Attune Fixed Bearing Posterior Stabilized total knee arthroplasty evaluated with KOOS. A prospective longitudinal cohort study with repetitive measurements 6 weeks, 3, 6, 12 and 24 months postoperative.

DETAILED DESCRIPTION:
Total knee arthroplasty is a well documented and efficient treatment method for degenerative knee arthritis. Nevertheless it is reported that 15-20% of patients are not satisfied with the result. Some of the complaints are anterior knee pain, mid flexion instability and range of motion. Attune Fixed Bearing Posterior Stabilized knee have been developed to address the common complaints after knee arthroplasty surgery . The investigators like to use the Attune Fixed Bearing Posterior Stabilized knee with patella resurfacing on 65 of Our departments eligible patients to evaluate the functional results. Our primary outcome measure is change in Knee Osteoarthritis Outcome Score.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 50-80 years eligible for total knee arthroplasty at our hospital

Exclusion Criteria:

* Patients unable to cooperate
* Larger deformity that not suitable for a Posterior Stabilized total knee prostheses.
* Revision operation
* Diagnosed with inflammatory arthritis
* Previously septic arthritis in the current knee joint
* Local malignancy/general bone metastases
* Serious Medical conditions that inflict on the walking ability
* Active infections, latent infections og increased risk og infection
* Previously arthrodeses or not well functioned arthroplasties in hips, knees or ankles.
* Neurologic illness with symptoms from the current limb

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score - (KOOS) | 2 years postoperative
  Knee injury and Osteoarthritis Outcome Score

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS-12) | 2 years postoperative
  Forgotten Joint Score -12. Translated Norwegian version
Quality of Life (EQ-5D) | 2 years postoperative
  Quality of life questionnaire
University of California Los Angeles-Activity score | 2 years postoperative
  Record change in Activity level
Range of Movement (ROM) | 2 years postoperative
  Range of movement pre- and postoperative
Stair climbing test functional test | 2 years postoperative
  Time spend on walking up and down 9 stairs
30 seconds stand up functional test | 2 years postoperative
  Number of stand ups from a chair in 30 seconds
40 meters walking functional test | 2 years postoperative
  Time spend on walking 40 meters
Visual Analogue Scale Satisfaction (VAS-satisfaction) | 2 years postoperative
  Scale for assesment of the satisfaction with the arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken HT, Baerum Hospital, Department of Medical Research, Sandvika, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Undecided